CLINICAL TRIAL: NCT00757055
Title: If Channel Blockade With Ivabradine in Patients With Diastolic Heart Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty recruit pts with PSHF HR > 70 & high BNP.
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dermot McCaffrey, Principal investigator, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N2008/Iva/DD
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Diastolic Heart Failure
Keywords: Heart failure; Diastolic heart failure; Heart failure with preserved systolic function; Heart failure with normal ejection fraction; Ivabradine; Diastolic dysfunction
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients on ivabradine titrated to heart rate
  Interventions: Drug: Ivabradine
- 2 (Placebo Comparator): No therapy given
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivabradine — Ivabradine titrated to heart rate starting at 5 mg bd and increasing to maximum of 7.5 mg bd or reducing to 2.5 mg if heart rate < 60 bpm.
  Other Names: Procoralen is brand name for Ivabradine
  Arms: 1
Drug: Placebo — No active treatment given
  Arms: 2

SUMMARY:
The purpose of this study is to investigate whether the medicine ivabradine, a novel drug which slows the heart rate has a favourable effect on patients with diastolic heart failure.

Ivabradine is a specific heart rate-lowering agent. It has a licence for treating patients with angina who are intolerant of agents such as beta blockers or whose angina is not adequately controlled. It has been shown to prolong exercise tolerance in these patients and to reduce the frequency of chest pain. Its mechanism of action is felt to be purely due to reducing heart rate, by as much as 10 beats per minute at rest, as well as by reducing the heart rate response to exercise.

Patients with diastolic heart failure often complain of breathlessness on exertion which relates to the stiffness or lack of compliance of their heart i.e. the heart fails to relax rapidly enough to allow it to fill with blood between each heart beat. This may result in high pressure in the heart chamber which backs up in to the lungs and may be experienced as breathlessness. There is little evidence that any specific therapy benefits patients with this type of heart failure besides treating coexisting problems such as high blood pressure or angina. By slowing the heart rate down with ivabradine, the heart would have a longer time to fill during exercise which would make it more effective. This slowing of the heart rate may therefore relieve the breathlessness experienced on activity such as walking to the shops or up a flight of stairs etc.

DETAILED DESCRIPTION:
Background:

Almost half of all patients with heart failure (HF) have preserved systolic function (PSHF) or heart failure with normal ejection fraction (HFNEF). Some of these have valvular abnormalities such as severe mitral or aortic regurgitation, severe anaemia, thyrotoxicosis or rarer tropical causes for heart failure. However, the majority of those with PSHF often have echocardiographic evidence of impaired diastolic function i.e. impaired relaxation and increased stiffness. This diastolic dysfunction may be related to age, hypertension or ischaemia. There is little evidence for any effective therapy in this large HF population despite randomised trials comparing placebo to ACE inhibitors i.e. perindopril in PEP-HF or angiotensin receptor blockers i.e. candesartan in the CHARM Preserved trial. There are also ongoing studies of aldosterone antagonists in diastolic heart failure i.e. eplerenone vs placebo in TOPCAT which continues to recruit.

In the absence of a strong evidence base, many physicians treat these patients with drugs that slow the heart rate, namely the calcium channel blocker verapamil and beta blockers. This has the effect of prolonging diastole or filling time and theoretically improving stroke volume thus reducing left ventricular end diastolic pressures (LVEDP) with resultant drop in wall stress and therefore less stimulus for myocardial fibrosis which exacerbates diastolic dysfunction by impeding compliance.

Hypothesis:

An alternative mechanism for slowing the heart rate is with ivabradine, a novel If channel blocker which acts purely on the sino atrial node with a mean heart rate lowering of 10 bpm in angina patients. This may result in improved diastolic filling which could be demonstrate by echocardiography, lower pulmonary capillary wedge pressures, which could be determined by measuring the E:E' ratio using tissue Doppler techniques, improving effort tolerance, estimated by assessing change in distance walked over 6 minutes and both a physician assessment using NYHA score as well as a patient Global Assessment and possibly better quality of life, determined by the Minnesota Living with Heart Failure Questionnaires.

Other theoretical improvements could be in the degree of stiffness or fibrosis due to reduced LV wall stress secondary to the longer filling time. This could be assessed using surrogates of wall strain such as brain natruretic peptide (BNP), wall stress as measured by strain rate imaging on echocardiography.

ELIGIBILITY:
Inclusion Criteria:

All patients must have a clinical diagnosis of diastolic heart failure as defined by all 3 of the following criteria:

* Presence of clinical heart failure for greater than or equal to 3 months before the screening visit. At the time of enrollment they should be in NYHA functional class I-III heart failure
* Left ventricular ejection fraction (LVEF) of greater than or equal to 50% (by echo or ventriculography) within 3 months of screening and LVEF still greater than or equal to 50% on day of enrollment
* BNP (b-type natruretic peptide) greater than or equal to 200 pg/ml at time of heart failure diagnosis
* Patients must be euvolaemic on clinical examination and have been clinically stable for at least 4 weeks with no medication changes
* Systolic blood pressure less than or equal to 150 mmHg but > 85 mmHg and diastolic blood pressure less than or equal to 95 mmHg for 4 weeks prior to and at the time of enrollment
* Able to walk at least 50 meters at time of enrollment

Exclusion Criteria:

* Aged < 18 or > 85
* Primary hemodynamically significant uncorrected valvular heart disease, obstructive or regurgitant
* Any planned revascularisation i.e. CABG or stenting or performed within last 90 days
* Any myocardial infarct within last 90 days
* Significant chronic obstructive airways disease in the opinion of the investigator
* Known infiltrative or hypertrophic obstructive cardiomyopathy or known pericardial constriction
* Inability to sign informed consent
* Atrial fibrillation
* Heart transplant recipient
* Currently implanted left ventricular assist device
* Stroke in past 90 days
* Gastrointestinal disorder that could interfere with study drug absorption
* Known intolerance to ivabradine
* Current participation (including prior 30 days) in any other therapeutic trial
* Any condition that, in the opinion of the investigator, may prevent the participant from adhering to the trial protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in echocardiographic indices of diastolic dysfunction | 12 weeks

SECONDARY OUTCOMES:
Improvement in 6 minute walk test | 12 weeks
Patient global assessment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dermot J McCaffrey, MB MRCPI FRACP, Principal Investigator — St Vincents University Hospital, Elm Park Dublin 4 Ireland
Locations (1):
- Heart Failure Unit, St Michaels Hospital, Dublin, Ireland